CLINICAL TRIAL: NCT00236756
Title: A Double-Blind Trial of Topiramate in Subjects With Lennox-Gastaut Syndrome.
Brief Title: A Study of the Efficacy and Safety of Topiramate as an add-on Therapy in the Treatment of Epilepsy Patients With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005464
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy; Seizures; Topiramate; Prophylaxis; Antiepileptic; Lennox-Gastaut syndrome; Seizures, tonic
MeSH Terms: conditions — Epilepsy; Seizures; Lennox Gastaut Syndrome | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of topiramate as add-on therapy in the treatment of epilepsy patients with Lennox-Gastaut syndrome, a severe form of epilepsy in which there are mixed types of seizures.

DETAILED DESCRIPTION:
Lennox-Gastaut syndrome is a severe form of epilepsy that usually develops in children 4 years of age and younger. It is characterized by several seizure types and developmental delay. Tonic seizures, in which the muscle tone is greatly increased and body, arms and legs make sudden stiffening movements, is particularly common in Lennox-Gastaut syndrome. Although atonic seizures, in which there is a sudden loss of muscle tone and strength, can occur in individuals with this syndrome. Control of seizures is difficult because they are usually resistant to antiepileptic drugs. Topiramate is a drug that is currently widely used for the treatment of seizures in adults and pediatric patients (2 to 16 years of age). This is a randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy and safety of topiramate as an add-on therapy in patients with Lennox-Gastaut syndrome. The study is composed of two phases: baseline (28 days) and double-blind treatment (approximately 11 weeks). Patients or their guardians/parents are given diaries to record information on seizures occurring during the study. During the baseline phase, the patient continues to receive the antiepileptic drug they have been taking. The double-blind phase is divided into two periods: titration, in which the topiramate dose was gradually increased (21 days) (patient's antiepileptic drug continues; this dose remains the same) and maintenance (56 days). The dose of both topiramate and the patient's antiepileptic drug remain constant during the maintenance period. Based on the investigator's judgment, all patients completing the double-blind period could be enrolled into an extension phase of the study. The primary assessment of effectiveness is the percent reduction from baseline in seizure rates (all types of seizures) in the double-blind phase. Safety assessments include the frequency of adverse events, results of clinical laboratory tests (hematology, biochemistry, and urinalysis), measurements of vital signs and body weight, physical examination and electrocardiogram findings, and neurological examinations. The study hypothesis is that topiramate is superior to placebo in reducing the seizure rate from baseline in the double blind phase of the study and is well tolerated. Topiramate (25milligram [mg] or 100mg tablets) or placebo, taken by mouth, starting at a dose of 1mg/kilogram(kg)/day, gradually increasing over 3 weeks to a total dose of 6mg/kg/day (given twice daily in equal oral doses for 8 weeks). Maximum daily dose is <=600mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 25 pounds
* diagnosis of Lennox-Gastaut syndrome and an electroencephalogram (EEG) with an abnormal pulsation pattern
* atypical absence seizures and drop attacks (i.e., tonic-atonic seizures) among other seizure types that could include tonic-clonic, myoclonic, and minor-motor
* at least 60 seizures during the month before baseline
* must be maintained on 1 or 2 antiepileptic drugs
* females must not have had their first menstrual period, or are physically incapable of child bearing, or if of child bearing potential, sexually abstinent, or using adequate contraceptive measures, and have a negative pregnancy test before study entry.

Exclusion Criteria:

* Patients whose seizures are due to a progressive disease (for example, active infection, cancer or metabolic disturbance)
* have a significant recent history (within 2 years) of medical diseases (respiratory, heart, gastrointestinal, blood diseases, rheumatic fever or cancer)
* history of alcohol or drug abuse.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 1993-08; Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in seizure rates (all types of seizures) in the double-blind phase. Percent reduction in drop attacks (tonic-clonic) and parent/guardian global evaluation at end of study

SECONDARY OUTCOMES:
Percent treatment responders all types of seizures. Percent treatment responders drop attacks (tonic-clonic seizures). Safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Sachdeo RC, Glauser TA, Ritter F, Reife R, Lim P, Pledger G. A double-blind, randomized trial of topiramate in Lennox-Gastaut syndrome. Topiramate YL Study Group. Neurology. 1999 Jun 10;52(9):1882-7. doi: 10.1212/wnl.52.9.1882. PMID 10371538
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- See also: A study of the efficacy and safety of topiramate in patients with Lennox-Gastaut syndrome — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=647&filename=CR005464_CSR.pdf